CLINICAL TRIAL: NCT06381661
Title: PALETTE- Adaptive Platform Trial for Personnalisation of Sepsis Treatment in Children and Adults: a Multi-national, Treatable Traits-guided, Adaptive, Exploratory, Bayesian Basket Trial
Brief Title: Adaptive Platform Trial for Personnalisation of Sepsis Treatment in Children and Adults: a Multi-national, Treatable Traits-guided, Adaptive, Exploratory, Bayesian Basket Trial
Acronym: PALETTE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP240385
Record Dates: First submitted 2024-04-09; First posted 2024-04-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
Keywords: Sepsis; Platform trial; Precision Medicine
MeSH Terms: conditions — Sepsis | interventions — tocilizumab; baricitinib; Interleukin 1 Receptor Antagonist Protein; Hydrocortisone; Fludrocortisone; Heparin; Heparin, Low-Molecular-Weight; sivelestat; interferon gamma-1b; Plasminogen

STUDY DESIGN:
Intervention Model Description: Randomization will concern 6 specific treatable traits (hyperinflammation, hypoinflammation, Macrophage Activation Like Syndrome, Corticoid response, hypercoagulation, Hypofibrinolysis). In each treatable trait, patients will be randomly allocated between control (usual care) and 1 to 4 experimental treatments using parallell arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- Hyperinflammation : Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab
- Hyperinflammation: Baricitinib (Experimental)
  Interventions: Drug: Baricitinib
- Hyperinflammation: Anakinra (Experimental)
  Interventions: Drug: Anakinra
- Hyperinflammation : blood purification with MTx.100 Plasma Adsorption Column (Experimental)
  Interventions: Other: blood purification with MTx.100 Plasma Adsorption Column
- Hyperinflammation : usual care (Active Comparator)
  Interventions: Other: Usual care
- Hypoinflammation : G CSF filgrastim (Experimental)
  Interventions: Drug: Heparin; Drug: G-CSF filgrastim
- Hypoinflammation : Interferon gamma-1b (Experimental)
  Interventions: Drug: Interferon gamma-1b
- Hypoinflammation : usual care (Active Comparator)
  Interventions: Other: Usual care
- MALS : Anakinra (Experimental)
  Interventions: Drug: Anakinra
- MALS : blood purification with MTx.100 Plasma Adsorption Column (Experimental)
  Interventions: Other: blood purification with MTx.100 Plasma Adsorption Column
- MALS : usual care (Active Comparator)
  Interventions: Other: Usual care
- Corticoids response : Hydrocortisone (Experimental)
  Interventions: Drug: Hydrocortisone
- Corticoids response : Fludrocortisone (Experimental)
  Interventions: Drug: Fludrocortisone
- Corticoids response : Hydrocortisone + Fludrocortisone (Experimental)
  Interventions: Drug: Hydrocortisone and fludrocortisone
- Corticoids response : usual care (Active Comparator)
  Interventions: Other: Usual care
- Hypercoagulation : Prophylactic unfractionated heparin (UFH) (Experimental)
  Interventions: Drug: Prophylactic unfractionated heparin (UFH)
- Hypercoagulation : Therapeutic UFH (Experimental)
  Interventions: Drug: Heparin
- Hypercoagulation : Therapeutic low molecular weight heparin (LMWH) (Experimental)
  Interventions: Drug: Low molecular weight heparin
- Hypercoagulation : Thrombomodulin (Experimental)
  Interventions: Drug: Recombinant humanThrombomodulin( rhTM)
- Hypercoagulation : usual care (Active Comparator)
  Interventions: Other: Usual care
- Hypofrinolysis : Sivelestat (Experimental)
  Interventions: Drug: Sivelestat
- Hypofrinolysis : OctaplasLG (Experimental)
  Interventions: Drug: Octaplas LG
- Hypofrinolysis : Plasminogen (Experimental)
  Interventions: Drug: Plasminogen
- Hypofrinolysis : Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Tocilizumab — 8 mg per kilogram of body weight enterally (oral or via a gastric tube) once daily for 14 days (or hospital discharge pending which will occur first) (same for adults and children)
  Arms: Hyperinflammation : Tocilizumab
Drug: Baricitinib — 4mg, enterally (oral or via a gastric tube) once daily for 14 days (or hospital discharge pending which will occur first) (same for adults and children)
  Arms: Hyperinflammation: Baricitinib
Drug: Anakinra — 100 mg subcutaneously once daily for 10 days (or hospital discharge pending which will occur first) (same for adults and children)
  Arms: Hyperinflammation: Anakinra; MALS : Anakinra
Drug: Hydrocortisone — 50mg (in children: 1-2 mg/kg) IV Q6 for 7 days
  Arms: Corticoids response : Hydrocortisone
Drug: Hydrocortisone and fludrocortisone — Hydrocortisone 50mg IV Q6 for 7 days + Fludrocortisone 50mg orally or via gastric tube once a day for 7 days.
  Arms: Corticoids response : Hydrocortisone + Fludrocortisone
Drug: Heparin — Therapeutic unfractionated heparin (UFH) starting at 400 (in children: 20 IU/kg/h) IU/kg/24h (target between 0.3 and 0.5 IU/ml), adapted to the therapeutic Partial Thromboplastin Time targeting values in the range of 60 to 100 seconds, with lower intensity dosing in the range of 60 to 80 seconds, for 7 days (or ICU discharge, pending which will occur first).
  Arms: Hypercoagulation : Therapeutic UFH; Hypoinflammation : G CSF filgrastim
Drug: Low molecular weight heparin — Therapeutic low weight molecular heparin (LMWH) tinzaparin, considering its contraindications, recommended dose ranges and monitoring if applicable, as follows: 175 (in children 100 U/kg) IU/kg/24h, for 7 days (or hospital discharge pending which will occur first).
  Arms: Hypercoagulation : Therapeutic low molecular weight heparin (LMWH)
Drug: Recombinant humanThrombomodulin( rhTM) — Recombinant human thrombomodulin (rhTM) 0.06 mg/kg/j IV, for 7 days (or ICU discharge, pending which will occur first).
  Arms: Hypercoagulation : Thrombomodulin
Drug: Sivelestat — 0.2 mg/kg/h for 7 days (or ICU discharge, pending which will occur first)
  Arms: Hypofrinolysis : Sivelestat
Other: Usual care — Usual care
  Arms: Corticoids response : usual care; Hypercoagulation : usual care; Hyperinflammation : usual care; Hypofrinolysis : Usual care; Hypoinflammation : usual care; MALS : usual care
Other: blood purification with MTx.100 Plasma Adsorption Column — up to 4 hours a day, up to four days in a row
  Arms: Hyperinflammation : blood purification with MTx.100 Plasma Adsorption Column; MALS : blood purification with MTx.100 Plasma Adsorption Column
Drug: G-CSF filgrastim — 0.5 MIU (5μg)/kg/day subcutaneously for 5 consecutive days (or up to ICU discharge pending which occurs first) - same for adults and children .
  Arms: Hypoinflammation : G CSF filgrastim
Drug: Interferon gamma-1b — rhIFNg subcutaneously at 50 µg/m2 if body surface >0,5 m2, or 1.5µg/kg if body surface of 0,5 m2or less, every other day for 15 days (or up to ICU discharge pending which occurs first)
  Arms: Hypoinflammation : Interferon gamma-1b
Drug: Fludrocortisone — 50µg orally (or via the gastric tube) once a day for 7 days (or ICU discharge pending which will occur first) (same for adults and children)
  Arms: Corticoids response : Fludrocortisone
Drug: Prophylactic unfractionated heparin (UFH) — 100 IU/kg/24h for 6 days
  Arms: Hypercoagulation : Prophylactic unfractionated heparin (UFH)
Drug: Octaplas LG — 12 mL/kg on day 1; repeated daily from day 2 to day 5, provided that PT/INR remains ≥ 1.40 (This intervention will be opened for randomisation once a supply circuit is in place)
  Arms: Hypofrinolysis : OctaplasLG
Drug: Plasminogen — 2,2 mg/kg/day (intravenous infusion) during 3 days.
  Arms: Hypofrinolysis : Plasminogen

SUMMARY:
PALETTE is a perpetual adaptive platform to efficiently study sepsis interventions within 'treatable traits' in all-ages patients enabling prompt evaluation of pandemic treatments. Treatable traits, therapeutic targets identified by phenotypes or endotypes (defined by biological mechanism or by treatment response) through validated biomarkers (measurable characteristic reflecting normal or pathogenic processes, or treatment responses), may include multi-omics, cellular, immune, metabolic, endocrine features, or intelligent algorithms. PALETTE Bayesian adaptive design enables parallel investigations of multiple interventions for sepsis, and quick inclusion of pandemic pathogens. PALETTE's new conceptual model will respond to the challenges of standard approaches, i.e. series of sepsis trials, each investigating one or two interventions, expensive, time consuming, and inappropriate in pandemic context.

ELIGIBILITY:
Platform inclusion criteria will be:

* All genders patients
* Aged >37 weeks corrected gestational age
* Sepsis as per Sepsis-3 definition for adults, and as per the PHOENIX sepsis for children

Briefly, all following criteria will be required:

1. Documented or suspected infection,
2. Sequential Organ Failure Assessment (SOFA) score ≥2 for adults, and PHOENIX sepsis score of ≥2 for children.

   * Health insurance

Platform exclusion criteria:

Any of the following:

* Refusal to consent for participating in the study,
* Pregnancy measured by beta-HCG blood levels
* Breast feeding
* Acute coronary disease in the past 3 months
* Stroke episode in the past 3 months
* Any condition for which patient's primary physician will consider inappropriate enrolling patient in the study

Treatable trait inclusion criteria :

* Hyperinflammation : Subphenotypes Beta, Delta, Gamma for adults; Subphenotypes PedSep-B, C, D for children
* Hypoinflammation : lymphocytes count < 1.0 × 10^9/L
* Macrophage Activation Like Syndrome : Ferritin >4,420 ng/mL for adults, Ferritin >500 ng/mL for children
* Corticosteroids: Positive for i-RECORDS algorithm signature
* Hypercoagulation (adults) : Prothrombin time (PT)/INR ≥ 1.40 AND Platelet count < 150 000/mm3 or greater than 30% decrease in platelets in 24 hours
* Hypofibrinolysis (adults): Plasminogen deficit < 0.5 µmol/L

There are also inclusion and exclusion criteria related to treatable traits and interventions.

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | At day 28
  Dual primary endpoint
Number of days alive without persistent life-supportive therapies | At day 28
  Dual primary endpoint Respiratory support: high flow oxygen, non-invasive or invasive mechanical ventilation, extracorporeal membrane oxygenation or CO2 removal; cardiovascular support: continuous infusion of any dose of vasopressor or inotrope, or mechanical circulatory assistance; renal support: intermittent or continuous renal replacement therapy

SECONDARY OUTCOMES:
Net benefit probability of intervention vs. control, assessed with a Generalized Pairwise Comparison (mortality prioritized over life-support-free days) | At day 28
  The Generalized Pairwise Comparison (GPC) method will be used to derive a single composite outcome. Each patient in the intervention group will be compared to each patient in the control group. For each pair, a score of +1, -1, or 0 will be assigned according to prioritized outcomes: (1) all-cause mortality at day 28, and (2) number of days alive without life-supportive therapies at day 28 if both patients have the same mortality status. The net benefit will be calculated as the sum of all pairwise scores divided by the total number of pairs, corresponding to the probability that a randomly chosen patient has a better outcome in one group than in the other.
Overall Survival | At day 90
Overall Survival | At 1 year
Overall Survival | At 3 years
Number of hospital free days | At 1 year
Number of hospital free days | At 3 years
Time to recover walking | At day 90
Time to resume previous social and professional activities | At 1 year
Quality of life score for adults assessed by SF-36 | At day 90
  The Short Form (36) (SF-36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Quality of life score for adults assessed by EQ-5D-5L | At day 90
  EQ-5D-5L : It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
Pediatric Quality of Life Inventory (PedsQL) | At day 90
  Standardized tool used to measure health-related quality of life (HRQoL) in children and adolescents (ages 2-18) It is a 23-item score divided in four domains : Phtsical functioning, Emotional functioning, Social functioning, School functioning The total score vary from 0 to 100. The higher the score the hiher the quality of life.
Quality of life score for children assessed by FSS | At day 90
  Functional Status Scale (FFS) : It examines 6 domains of functioning, and each domain receives a score of 1 (normal), 2 (mild dysfunction), 3 (moderate dysfunction), 4 (severe dysfunction), or 5 (very severe dysfunction). Final scores range from 6 to 30.
Quality of life score for adults assessed by SF-36 | At 1 year
  The Short Form (36) (SF-36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Quality of life score for adults assessed by EQ-5D-5L | At 1 year
  EQ-5D-5L : It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
Quality of life score for children assessed by FSS | At 1 year
  Functional Status Scale (FFS) : It examines 6 domains of functioning, and each domain receives a score of 1 (normal), 2 (mild dysfunction), 3 (moderate dysfunction), 4 (severe dysfunction), or 5 (very severe dysfunction). Final scores range from 6 to 30.
Pediatric Quality of Life Inventory (PedsQL) | At 1 year
  Standardized tool used to measure health-related quality of life (HRQoL) in children and adolescents (ages 2-18) It is a 23-item score divided in four domains : Phtsical functioning, Emotional functioning, Social functioning, School functioning The total score vary from 0 to 100. The higher the score the hiher the quality of life.
Quality of life score for adults assessed by SF-36 | At 3 years
  The Short Form (36) (SF-36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
  Ware JE, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. Conceptual framework and item selection. Med Care 1992;30:473-83.
Quality of life score for adults assessed by EQ-5D-5L | At 3 years
  EQ-5D-5L : It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
Quality of life score for children assessed by FSS | At 3 years
  Functional Status Scale (FFS) : It examines 6 domains of functioning, and each domain receives a score of 1 (normal), 2 (mild dysfunction), 3 (moderate dysfunction), 4 (severe dysfunction), or 5 (very severe dysfunction). Final scores range from 6 to 30.
Pediatric Quality of Life Inventory (PedsQL) | At 3 years
  Standardized tool used to measure health-related quality of life (HRQoL) in children and adolescents (ages 2-18) It is a 23-item score divided in four domains : Phtsical functioning, Emotional functioning, Social functioning, School functioning The total score vary from 0 to 100. The higher the score the hiher the quality of life.
Number of adverse events | Up to 3 years
  Tolerance of interventions considering any grade of 3 serious adverse events.
Incidence of new sepsis episodes | At day 90
Incidence of new sepsis episodes | At 1 year
Incidence of new sepsis episodes | At 3 years
Incidence of new unscheduled hospitalizations | At day 90
Incidence of new unscheduled hospitalizations | At 1 year
Incidence of new unscheduled hospitalizations | At 3 years
Incidence of sequels in neurocognitive, neuromuscular; cardiovascular, respiratory, renal, metabolic, and immune systems | At 3 years
Number of grade 3 serious adverse events | At day 28

OTHER OUTCOMES:
Circulating levels of cytokines | At inclusion
Circulating levels of chemokines | At inclusion
Circulating levels of cytokines | At day 1
Circulating levels of chemokines | At day 1
Circulating levels of cytokines | At day 7
Circulating levels of chemokines | At day 7
Circulating levels of cytokines | At 1 year
Circulating levels of chemokines | At 1 year
Circulating levels of cytokines | At 3 years
Circulating levels of chemokines | At 3 years

IPD SHARING:
Plan to Share IPD: Undecided